CLINICAL TRIAL: NCT06772792
Title: A Clinical Study to Evaluate the Effect of MK-0616 on the Pharmacokinetics of Alendronate in Healthy Adult Participants
Brief Title: A Study to Evaluate the Drug-Drug Interaction Between Enlicitide Decanoate (MK-0616) and Alendronate in Healthy Adult Participants (MK-0616-027)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-027; MK-0616-027 (Other: MSD)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Alendronate; MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alendronate (Experimental): Participants receive a single oral dose of alendronate on Day 1 OR participants receive a single oral dose of alendronate on Day 15 depending on randomization.
  Interventions: Drug: Alendronate
- Alendronate + Enlicitide Decanoate (Experimental): Participants receive an oral dose of alendronate plus an oral dose of enlicitide decanoate on Day 1 OR participants receive an oral dose of alendronate plus an oral dose of enlicitide decanoate on Day 15 depending on randomization.
  Interventions: Drug: Alendronate; Drug: Enlicitide Decanoate

INTERVENTIONS:
Drug: Alendronate — Oral administration
  Other Names: Fosamax®
Drug: Enlicitide Decanoate — Oral administration
  Other Names: MK-0616
  Arms: Alendronate + Enlicitide Decanoate

SUMMARY:
The goal of this study is to learn what happens to a single dose of alendronate over time in a healthy participant's body when the participant is given a single dose of enlicitide decanoate. Researchers want to learn how safe and tolerable is the co-administration of enlicitide decanoate and alendronate.

ELIGIBILITY:
Inclusion Criteria:

* Has no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and electrocardiograms (ECGs)
* Has a body mass index (BMI) ≥18.0 kg/m^2 and ≤32.0 kg/m^2 (inclusive)

Exclusion Criteria:

* Has a history or presence of abnormalities of the esophagus which delay emptying such as stricture or achalasia
* Has a history of cancer (malignancy)
* Has a history of gastrointestinal disease which may affect food and drug absorption

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine the AUC0-Last of alendronate.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine the AUC0-Inf of alendronate.
Maximum Plasma Concentration (Cmax) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine the Cmax of alendronate.
Time to Maximum Plasma Concentration (Tmax) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine the Tmax of alendronate.
Apparent Terminal Half-Life (t1/2) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine the t1/2 of alendronate.
Apparent Clearance (CL/F) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine the CL/F of alendronate.
Apparent Volume of Distribution (Vz/F) of Alendronate | At designated timepoints (up to approximately 10 hours post-dose)
  Blood samples will be collected to determine Vz/F of alendronate.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 3 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.
Total Amount of Alendronate Excreted Unchanged Over a Period of 48 Hours (Ae0-48) after Alendronate Administration | At designated timepoints (up to approximately 48 hours post-dose)
  Urine samples will be collected to determine the Ae0-48 of alendronate.
Maximum Rate (Rmax) of Alendronate Excretion | At designated timepoints (up to approximately 48 hours post-dose)
  Urine samples will be collected to determine the Rmax of alendronate excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com